CLINICAL TRIAL: NCT06084858
Title: Effect of Dialysate Bicarbonate Prescription on Serum Calcification Propensity and Calciprotein Particles in Hemodialysis Patients
Brief Title: Effect of Changes in Dialysate Bicarbonate on Serum Calcification Propensity and Calciprotein Particles in Hemodialysis Patients
Acronym: D-Bic-T50-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Priv. Doz. Dr. Daniel Cejka (Other)
Responsible Party: Sponsor-Investigator, Prim. Priv. Doz. Dr. Daniel Cejka, Principal Investigator, Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: D-Bic-T50-HD
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, proof-of-priciple, pilot study. Bicarbonate for dialysis will be modified step-by-step from 27 mmol/l to 37 mmol/l.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialysate Bicarbonat modification (Experimental): Dialysate bicarbonate prescription will be modified from low (27 mmol/l) to high (37 mmol/l) in a step-wise fashion
  Interventions: Other: Dialysate bicarbonate modification

INTERVENTIONS:
Other: Dialysate bicarbonate modification — Dialysate bicarbonate prescription will be modified from low (27 mmol/l) to high (37 mmol/l) in a step-wise fashion

SUMMARY:
This is a single-center, prospective, proof-of-priciple, pilot study in 24 end-stage renal disease patients on chronic hemodiaysis.

DETAILED DESCRIPTION:
This single-arm, proof-of-principle study will be conducted at the dialysis facility of the Ordensklinikum Linz Elisabethinen Hospital. The dialysate bicarbonate prescription will be decreased from standard of care (usually 35mmol/l) in a stepwise fashion (2 mmol/l per change) to 27 mmol/l and subsequentially increased in a stepwise fashion (2 mmol/l per change) to 37 mmol/l over the course of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* chronic (≥3 months) treatment with hemodialysis or hemodiafiltration
* stable clinical condition

Exclusion Criteria:

* inability to provide informed consent
* dialysis treatment less than thrice weekly
* morbid obesity (body mass index >40 kg/m2)
* chronic inflammation (C reactive protein >10 mg/dL, reference: <0.5 g/dL)
* current immunosuppressive medication,
* severe chronic obstructive pulmonary disease (COPD stage III or IV)
* history of severe hypercapnia or hypoxemia
* overt congestive heart failure
* history of severe hypokalemia (<3.0 mmol/l) or hyperkalemia (>6.5 mmol/L) within 3 months prior to study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
T50-Laboratory Test for measuring calcification | 6 Weeks
  The intra-individual difference of T50-times between low (27 mmol/l) and high (37 mmol/l) dialysate bicarbonate prescription.

SECONDARY OUTCOMES:
CPP Levels | 6 Weeks
  The difference in intra-dialytic change in CPP levels with low (27 mmol/l) and high (37 mmol/l) dialysate bicarbonate prescription, while the inter-dialytic differences in CPP levels with low and high dialysate bicarbonate prescriptions will be tertiary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cejka, MD, Principal Investigator — Head of Nephrology
Locations (1):
- Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria, Austria